CLINICAL TRIAL: NCT07106190
Title: Evaluation of Secondary Complication Awareness Among Caregivers of Post-stroke Patients
Brief Title: Seconder Complication Awareness of Caregivers
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-20024-1193
Record Dates: First submitted 2025-07-07; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Stroke Rehabilitation
Keywords: Stroke Rehabilitation; Seconder Complications; Caregiver awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers who stay patient more than one month
  Interventions: Other: Patients will be informed during the rehabilitation process

INTERVENTIONS:
Other: Patients will be informed during the rehabilitation process — Patients will be informed during the rehabilitation process about secondary complications of stroke

SUMMARY:
Stroke-related secondary complications increase the length of hospital stay, negatively affect the functional expectation in the rehabilitation process and increase repeated hospital admissions. For these reasons, complications secondary to stroke are associated with mortality and increased economic burden. Prevention of secondary complications is important. Increasing the level of knowledge and awareness of caregivers, who are constantly with the patient, about secondary complications is effective in preventing secondary complications. The aim of this study was to evaluate the level of awareness of caregivers about secondary complications related to stroke and the effect of rehabilitation process. There is no study or scale evaluating the level of awareness of secondary complications related to stroke in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Followed by ischaemic or haemorrhagic stroke
* No more than 1 year has passed since the date of the incident
* Followed with the same caregiver for at least 1 month
* Patients and carers over 18 years of age

Exclusion Criteria:

* Cognitive or psychological impairment of the caregiver
* Not volunteering to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers of post stroke patients who are hospitalised for rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Test | first day of hospitalisation and 4th week of hospitalisation
  The test will assess caregivers' level of knowledge about secondary complications. Secondary complications to be investigated include spasticity and joint contracture, dysphagia and aspiration, depression, hemiplegic shoulder, fall and fracture risk, central pain, neurogenic bladder and urinary tract infection, pressure ulcer, convulsion, deep vein thrombosis and pulmonary embolism. The test will consist of a total of 20 questions using true/false questions respectively. Patients can take points between 0 and 20. Higher points mean better results.

SECONDARY OUTCOMES:
The Questionnaire | First day of hospitalisation, 4th week of hospitalisation
  The questionnaire will assess caregivers' ideas about their level of knowledge about secondary complications. Secondary complications to be investigated include spasticity and joint contracture, dysphagia and aspiration, depression, hemiplegic shoulder, fall and fracture risk, central pain, neurogenic bladder and urinary tract infection, pressure ulcer, convulsion, deep vein thrombosis and pulmonary embolism. The questionnaire will consist of a total of 20 questions using10-point Likert scale respectively. Patients can take points between 0 and 200. Higher points mean better results.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)